CLINICAL TRIAL: NCT03637244
Title: Pilot Randomized Controlled Trial of a Decision Support Intervention Adapted for HIV Pre-Exposure Prophylaxis Adoption and Adherence Among African, Caribbean and Black Canadian Patients
Brief Title: Decision Support Intervention Adapted for HIV Pre-Exposure Prophylaxis for Adoption and Adherence for Black Canadians
Acronym: PrEPDSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: StMichaelnelsonla
Record Dates: First submitted 2018-01-22; First posted 2018-08-17 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: HIV/AIDS
Keywords: HIV PrEP Decision support African Caribbean Black Canadians
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: H1: PrEP decision support increases decision quality in both LDQ and HDQ groups, H2: HDQ + decision-support group more likely to initiate PrEP than HDQ control, H3: HDQ PrEP initiators are more likely than LDQ initiators to have serum levels consistent with adherence at 60-days. Investigators supply one smartphone/ participant,each registered to St. Mike's Hospital to protect participant privacy. The decision support aid will be a pre-programmed bookmark, an RA will give participants a brief tutorial on its use. Patients assigned to the experimental condition (LDQ + DS and HDQ + DS) will use the bookmarked link to the decision-aid within the first 7-14 days (and thereafter as needed) during the study period. The routine care group will be asked to use a bookmarked link to frequently asked questions on tenofovir + emtricitabine for PrEP. All groups will be compared on decision-quality at 14-days, self-reported PrEP initiation at 30-days, and PrEP adherence at 60-days post enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Condition (Experimental): Patients assigned to the experimental condition (LDQ + DS and HDQ + DS) will be asked to use the bookmarked link to the decision-aid within the first 7-14 days (and thereafter as needed) during the study period. The routine care group will be asked to use a bookmarked link to frequently asked questions on tenofovir + emtricitabine for PrEP. All groups will be compared on decision-quality at 14-days, self-reported PrEP initiation at 30-days, and PrEP adherence at 60-days post enrollment.
  Interventions: Behavioral: Decision Support Aid and PrEP for Black Canadians

INTERVENTIONS:
Behavioral: Decision Support Aid and PrEP for Black Canadians — Ottawa Decision Support Framework Adaptation.Investigators will use the inputs from the qualitative findings, CDC public health guidance and the tenofovir + emtricitabine product monograph to tailor the ODSF for use in the C5TM PrEP decision support web-app.

SUMMARY:
Aim 1: Adapt Ottawa Decision Support Framework for the HIV PrEP decisional needs of African, Caribbean and Black (ACB) Canadian patients Aim 2. Pilot Test The Adapted Decision-Support Intervention Using a Two-Arm Randomized Controlled Design

DETAILED DESCRIPTION:
Aim 1: Adapt Ottawa Decision Support Framework for the HIV PrEP decisional needs of ACB Canadian patients. Investigators propose a cross-sectional qualitative descriptive study using data collected from key informant interviews with PrEP eligible patients and surveys with health professionals involved in HIV PrEP management. Under this aim two research questions will be investigated.

Q1) What factors do ACB Canadian patients consider when deciding whether to adopt HIV PrEP? Q2. How do SDT constructs of autonomy, competence and relatedness influence ACB Canadian's decision-making experiences regarding PrEP adoption?

AIM 2. Pilot Test The Adapted Decision-Support Intervention Using a Two-Arm Randomized Controlled Design.Hypothesis testing will be de-emphasized in favor of generating effect size estimates. Under this aim three research questions will be investigated. Preliminary hypotheses include:

H1: PrEP decision support increases decision quality in both LDQ and HDQ groups, H2: HDQ + decision-support group more likely to initiate PrEP than HDQ control, H3: HDQ PrEP initiators are more likely than LDQ initiators to have serum levels consistent with adherence at 60-days.

Data on decision quality survey and PrEP initiation data will generated by the subject from self-administered assessments via the decision-support app on the study-issued smartphone. Investigators will also collect biological specimens to measure adherence to HIV PrEP at 60-days post enrollment.

The study will take place in the Toronto metropolitan area (pop. 2.5 million). Over half (59%) of Canada's ACB population is settled in the province of Ontario. Moreover, the majority (70%) of ACB people in Ontario live in metro Toronto, making it the ideal location for this study. The trial procedures will be conducted at sites within the St. Michael's Hospital (SMH) system, including the SMH Li Ka Shing Knowledge Institute.

ELIGIBILITY:
Inclusion Criteria

* Self identify as Black African, Caribbean and or Canadian
* HIV sero-negative
* Not in a monogamous sexual partnership with a recently tested HIV negative man
* Self report unprotected anal sex with a man in the past six months
* Diagnosed with gonorrhea, chlamydia or syphilis in the past six months
* Are in an ongoing sexual relationship with an HIV positive partner
* Currently live in the Greater Toronto metropolitan area
* Can speak and understand either English or French

Exclusion Criteria

* Non Black African Caribbean and or Canadian person
* Diagnosed with HIV and or AIDS
* Unable to consent to provide documentation of negative HIV status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men, women cisgender and transgender inclusive based on self representation
Enrollment: 90 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in baseline (initiation of PrEP) to adherence of PrEP for ACB Canadians | Self-reported PrEP initiation at 30-days and PrEP adherence at 60-days post enrollment.
  PrEP Initiation (does the person fill a prescription for PrEP) PrEP Adherence (analysis of intracellular tenofovir+emtricitabine concentration in dried blood spot)

CONTACTS AND LOCATIONS:
Overall Officials: LaRon E Nelson, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital Academic Family Health Team, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Study findings (no identifiable data is included) will be shared via study participant focused community meeting first. Then findings will be published in peer reviewed journals and other relevant publications